CLINICAL TRIAL: NCT00532168
Title: Once-daily Antiretroviral Therapy in HIV-1 Infected Patients With CD4+ Cell Counts Below 100 Cells/Mcl. A Prospective, Randomized, Multicentre, Open Clinical Study.
Brief Title: Once-daily Antiretroviral Therapy in HIV-1 Infected Patients With CD4+ Cell Counts Below 100 Cells/Mcl
Acronym: ADVANZ-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVANZ-3; EudraCT: 2006-006268-42; FIS grant: EC07/90642
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: advanced HIV-infected patients; late presenters; antiretroviral therapy; immune reconstitution; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; efavirenz; Lopinavir; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): tenofovir plus emtricitabine plus efavirenz
  Interventions: Drug: tenofovir + emtricitabine + efavirenz
- 2 (Experimental): tenofovir plus emtricitabine plus lopinavir-ritonavir
  Interventions: Drug: tenofovir + emtricitabine + lopinavir-ritonavir
- 3 (Experimental): tenofovir plus emtricitabine plus atazanavir-ritonavir
  Interventions: Drug: tenofovir + emtricitabine + atazanavir-ritonavir

INTERVENTIONS:
Drug: tenofovir + emtricitabine + efavirenz — tenofovir + emtricitabine + efavirenz, approved dose, oral route, QD
  Arms: 1
Drug: tenofovir + emtricitabine + lopinavir-ritonavir — tenofovir + emtricitabine (QD) + lopinavir-ritonavir (BID), oral route, approved dose
  Arms: 2
Drug: tenofovir + emtricitabine + atazanavir-ritonavir — tenofovir + emtricitabine + atazanavir + ritonavir (100 mg), oral route, approved dose, QD
  Arms: 3

SUMMARY:
There are few randomized clinical trials in advanced HIV patients. This is a multicenter, randomized, open clinical trial, comparing three parallel groups, to compare the immunological reconstitution and the virological efficacy and safety of three different combinations of antiretroviral therapy given once a day (QD): tenofovir plus emtricitabine plus either efavirenz, lopinavir-ritonavir or atazanavir-ritonavir during 96 weeks in advanced antiretroviral naïve HIV-1 infected patients with less than 100 CD4+ T-cells/mm3. Primary endpoint is the median increase in CD4+ T-cell count at 48 weeks after starting HAART.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV-1 infection
* Age 18 or more
* Antiretroviral-naive
* Baseline CD4+ count <100 cels/mcL.
* No mutations of drug resistance at baseline (M184V/I, K65R, resistance to efavirenz or 2 or more PRAMs (L33I/F/V, V82A/F/L/T, I84V, L90M)
* Written informed consent

Exclusion Criteria:

* Hypersensibility to study drugs.
* Pregnancy or breastfeeding
* Active OI requiring admission
* Active lymphoma or malignancy (Kaposi sarcoma included)
* Cl creatinine below 30 ml/min.
* Liver failure
* Treatment with nephrotoxic drugs, immunomodulators, interleukine-2, systemic steroids or investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Median increase in CD4+ T-cell count at 48 weeks after starting the HAART combination randomly assigned | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Miró, MD, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Miro JM, Manzardo C, Ferrer E, Lonca M, Guardo AC, Podzamczer D, Domingo P, Curran A, Clotet B, Cruceta A, Lozano F, Perez I, Plana M, Gatell JM; Advanz-3 Study Group. Immune Reconstitution in Severely Immunosuppressed Antiretroviral-Naive HIV-1-Infected Patients Starting Efavirenz, Lopinavir-Ritonavir, or Atazanavir-Ritonavir Plus Tenofovir/Emtricitabine: Final 48-Week Results (The Advanz-3 Trial). J Acquir Immune Defic Syndr. 2015 Jun 1;69(2):206-15. doi: 10.1097/QAI.0000000000000567. PMID 25831464